CLINICAL TRIAL: NCT01437722
Title: A Double-blind, Multicenter, Randomized, Placebo-controlled, Dose-ranging Study to Determine the Efficacy and Safety of SPL7013 Gel (VivaGel®) Administered Vaginally to Prevent the Recurrence of Bacterial Vaginosis
Brief Title: Dose-ranging Study of SPL7013 Gel for the Prevention of Bacterial Vaginosis (BV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPL7013-014
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Bacterial Vaginosis (BV)
Keywords: BV; Bacterial vaginosis; recurrent; SPL7013 Gel; VivaGel
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1% SPL7013 Gel (Experimental)
  Interventions: Drug: 1% SPL7013 Gel
- 3% SPL7013 Gel (Experimental)
  Interventions: Drug: 3% SPL7013 Gel
- placebo gel (Placebo Comparator)
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: 1% SPL7013 Gel — vaginal gel
  Arms: 1% SPL7013 Gel
Drug: 3% SPL7013 Gel — vaginal gel
  Arms: 3% SPL7013 Gel
Drug: placebo gel — vaginal gel
  Arms: placebo gel

SUMMARY:
The purpose in this clinical study is to determine the efficacy of SPL7013 Gel for the prevention of recurrence of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years with a history of recurrent BV, defined as at least 3 documented episodes in the previous 12 months (including the current episode).
* Current episode of BV as defined by subject-reported symptoms and Amsel's Criteria
* Otherwise healthy

Exclusion Criteria:

* No active STIs and/or current UTI
* Previous exposure to SPL7013 Gel
* A Papanicolaou (Pap) smear result considered to be clinically significant (ie, high grade cervical intraepithelial squamous lesions [HSIL] on cytology or cervical intraepithelial neoplasia [CIN] grades of CIN2 or CIN3 on histology) in the previous 2 years or in accordance with local treatment guidelines.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of women who have experienced a recurrent episode of BV as a measure of efficacy | Day 112 +/- 5
  Number of women who have BV as measured by subject-reported symptoms and Amsel's Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Paull, PhD, Study Director — Starpharma Pty Ltd